CLINICAL TRIAL: NCT01670162
Title: On-label tReatment With Intravitreal Aflibercept Injection for Patients With Persistent Pigment Epithelial Detachments in Neovascular AMD.
Brief Title: On-label tReatment With Intravitreal Aflibercept injectiOn for Patients With Persistent Pigment epitheliaL Detachments in Neovascular Age Related Macular Degeneration (AMD)
Acronym: ROLL
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tennessee Retina (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGFT-OD-1220
Record Dates: First submitted 2012-08-17; First posted 2012-08-21 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Age Related Macular Degeneration; Pigment Epithelial Detachment
Keywords: Pigment Epithelium of Eye; Wet macular degeneration; Macular degeneration
MeSH Terms: conditions — Macular Degeneration; Retinal Detachment; Wet Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3 loading doses, then every 2 months (Experimental): All patients will receive 3 monthly intravitreal aflibercept injections followed by mandatory dosing every 3 months. If needed, patients can be treated monthly.
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept — Intravitreal Injection 2mg/0.05mL Aflibercept
  Other Names: VEGF-Trap; Eylea

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of intravitreal aflibercept injection in a population of neovascular AMD patients that have been previously treated with 2.0 mg ranibizumab for persistent PEDs.

DETAILED DESCRIPTION:
A Phase 4 study to evaluate the efficacy and safety of intravitreal aflibercept injection in a population of neovascular AMD patients that have been previously treated with 2.0 mg ranibizumab for persistent PEDs (the ROLL study).

ELIGIBILITY:
Inclusion Criteria:

* Previous enrollment in the study evaluating 2.0mg ranibizumab (NCT 01189019) without early study discontinuation. The last treatment* in the study eye should have been received at least 30 days before enrollment in this study.

  **last study treatment of either 1.0mg or 2.0mg ranibizumab
* Presence of persistent fibrovascular pigment epithelial detachment Willing and able to comply iwth clinic visits and study related procedures Provide signed informed consent

Exclusion Criteria:

* Prior treatment with verteporfin, or external beam radiation therapy, or transpupillary thermotherapy in the study eye.

Previous subfoveal focal laser photocoagulation involving the foveal center in the study eye.

* History of vitrectomy, submacular surgery, or other surgical intervention for AMD in the study eye.
* Concurrent eye disease in the study eye that could compromise visual acuity (e.g. diabetic retinopathy, advanced glaucoma).
* Any concurrent intraocular condition in the study eye (e.g. diabetic retinopathy or glaucoma) that, in the opinion of the investigator, could either require medical or surgical intervention during the 12 month study period to prevent or treat visual loss that might result from that condition, or if allowed to progress untreated, could likely contribute to loss of at least 2 Snellen equivalent lines of best corrected visual acuity over the 12 month study period.
* Active intraocular inflammation (grade trace or above) in the study eye, or history of idiopathic or auto-immune associated uveitis in either eye.
* Current vitreous hemorrhage in the study eye.
* History of rhegmatogenous retinal detachment or macular hole (stage 3 or 4) in the study eye.
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye.
* Aphakia, anterior chamber intraocular lens (ACIOL) or unstable posterior chamber intraocular lens (PCIOL).
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure equal to or greater than 30 despite treatment with anti-glaucoma medication).
* Pregnant or breastfeeding women.
* Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraception measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device (IUD); bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam or jelly).

  * Contraception is not required for men with documented vasectomy. **Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-08; Primary Completion 2015-11 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with flattening of PED | 12 months

SECONDARY OUTCOMES:
Mean Change in Best Corrected Visual Acuity (BCVA) | 6 month timepoint and 12 month timepoints
Proportion of patients with flattening of PED | 6 months
Proportion of patients with flattening of PED | 18 month and 24 month timepoints
Mean number of injections needed | 12 month period
Mean change in Optical Coherence Tomography (OCT) central retinal thickness | 6 month and 12 month timepoints
Proportion of patients gaining 5 letters or more letters on Early Treatment Diabetic Retinopathy Study (ETDRS) Chart | 6 month and 12 month timepoint
Mean change in BCVA | 18 month and 24 month timepoint
Mean number of injections | during year 2
Mean change in OCT central retinal thickness | 18 month and 24 month timepoints
Proportion of patients gaining 5 letters or more | 18 month and 24 month timepoints

OTHER OUTCOMES:
Incidence and severity of adverse events | 24 month period

CONTACTS AND LOCATIONS:
Overall Officials: Brandon G Busbee, MD, Principal Investigator — Tennessee Retina, PC
Locations (3):
- United States (3):
  - Pacific Eye Associates, San Francisco, California
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Tennessee Retina, P.C., Nashville, Tennessee